CLINICAL TRIAL: NCT03809936
Title: Effects of Transcranial Direct Current Stimulation on the Disorders of Consciousness
Brief Title: Transcranial Direct Current Stimulation in Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS
Record Dates: First submitted 2018-07-26; First posted 2019-01-18 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2019-04

CONDITIONS: Disorder of Consciousness
Keywords: tDCS; EEG
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: Using a sham-controlled randomized double-blind design, 20 patients were randomly assigned to either a real or sham stimulation group. Each intervention week included 10 daily sessions of 20-minute therapy with either anodal transcranial direct current stimulation (2 mA, 20 minutes; experimental group) or sham transcranial direct current stimulation (control group) over the left dorsolateral prefrontal cortex (DLPFC).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Active Comparator): real tDCS:anodal transcranial direct current stimulation were delivered over the left DLPF cortex for 20 minutes in patients.
  Interventions: Device: real tDCS
- sham tDCS (Sham Comparator): sham tDCS:sham transcranial direct current stimulation were delivered over the left DLPF cortex for 20 minutes in patients.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: real tDCS — Direct current was applied by a battery-driven constant current stimulator using saline-soaked surface sponge electrodes (7 3 5 cm) with the anode positioned over the left dorsolateral prefrontal cortex (F3 according to the 10-20 international system for EEG placement) and the cathode placed over the right supraorbital region. During real tDCS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes.
  Arms: real tDCS
Device: sham tDCS — For the sham condition(sham tDCS), the same electrode placement was used as in the stimulation condition, but the current was applied for only 5 seconds, and was then ramped down.
  Arms: sham tDCS

SUMMARY:
To date, several studies have focused on the use of transcranial direct current stimulation(tDCS) in patients with impaired consciousness.However,its therapeutic effects have been variously documented.So,in this study ,investigators explore the effects of tDCS.

DETAILED DESCRIPTION:
Background:tDCS was supposed as an experimental approach to disorders of consciousness treatment. Its therapeutic effects have been variously documented.

Objective: The study aimed to investigate the reactivity of electroencephalography (EEG) and the clinical response of patients with disorders of consciousness and explore the neuromodulatory effects of highfrequency tDCS in DOC.

Method:In this double-blind, randomized controlled trial,real or sham tDCS were applied to the left dorsolateral prefrontal (DLPF) cortex of participants with disorders of consciousness for two weeeks. Evaluations were blindly performed at baseline, immediately after the end of the 14-days treatment and 1 week later with the JFK Coma Recovery Scale-Revised (CRS-R) scale and EEG.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of DOC
2. Ages 14 to 65 years old
3. No centrally acting drugs
4. No neuromuscular function blockers and no sedation within the prior 24 hours;

Exclusion Criteria:

1. History with nervous or spirit disorders, or some other serious diseases
2. A contraindication for tDCS

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the JFK Coma Recovery Scale-Revised (CRS-R) scale | at baseline (T0), immediately after the end of the treatment (T1), 1 week later (T2).Investigators observed the changes from baseline to the end of stimulation.
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.

SECONDARY OUTCOMES:
EEG data ( electrophysiological parameters) | at baseline (T0), immediately after the end of the treatment (T1), 1 week later (T2).
  delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz) and beta (12-30 Hz).an increase of delta and theta activity usually reflects encephalopathy and/or structural lesions, interpreted as poor outcome predictor of DOC .The power of α and β is related to the chance of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu J, Wu Y, Wu B, Xu C, Cai J, Wen X, Meng F, Zhang L, He F, Hong L, Gao J, Li J, Yu J, Luo B. Sleep patterns correlates with the efficacy of tDCS on post-stroke patients with prolonged disorders of consciousness. J Transl Med. 2022 Dec 15;20(1):601. doi: 10.1186/s12967-022-03710-2. PMID 36522680
- [Derived] Wu M, Yu Y, Luo L, Wu Y, Gao J, Ye X, Luo B. Efficiency of Repetitive Transcranial Direct Current Stimulation of the Dorsolateral Prefrontal Cortex in Disorders of Consciousness: A Randomized Sham-Controlled Study. Neural Plast. 2019 Jun 11;2019:7089543. doi: 10.1155/2019/7089543. eCollection 2019. PMID 31308848